CLINICAL TRIAL: NCT00241501
Title: A Phase III, Multicentre, Randomized, Double-blind, Parallel-group Study to Evaluate the Safety of Once Daily Esomeprazole for the Treatment of Clinically Diagnosed Gastroesophageal Reflux Disease (GERD) in Pediatric and Adolescent Patients 12 to 17 Years of Age, Inclusive.
Brief Title: Safety of Daily Dose Esomeprazole for GERD for Pediatric and Adolescent Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9614C00098
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole (Nexium)

SUMMARY:
This study is a phase III, multi-centre, randomized, double-blind study to assess the safety and tolerability of once daily treatment with esomeprazole 20 or 40 mg in pediatric and adolescent patients 12 to 17 years of age, inclusive, with clinically diagnosed GERD. The treatment period will be up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent from the patient's parent/guardian, and assent from the patient prior to conducting of any study-related procedures.
* Patients must be male or female between the age of 12 and 17 years, inclusive.
* Patients must have a clinical diagnosis of GERD made by the investigator based on any of the following factors: history, physical examination, review of systems, laboratory test results, or information from diagnostic testing.

Exclusion Criteria:

* Patients who have used a PPI within 14 days prior to randomization, including over-the-counter Prilosec®.
* Patients who have used any prescription or over-the-counter treatment for symptoms of gastroesophageal reflux disease (GERD), such as Histamine 2 Receptor Antagonists (H2RA) or prokinetics, within 3 days prior to randomization. Antacids may be used, except for those containing bismuth.
* Patients with a known hypersensitivity, allergy, or intolerance to any component of esomeprazole or omeprazole.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140
Dates: Start 2004-02; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To evaluate safety & how tolerable a once daily treatment with esomeprazole is in pediatric & adolescent patients
12 to 17 years of age, inclusive, with clinically diagnosed Gastroesophageal Reflux Disease (G

SECONDARY OUTCOMES:
To evaluate the clinical outcome of once daily treatment with esomeprazole in relieving gastroesophageal reflux disease (GERD)-associated signs & symptoms in pediatric & adolescent patients 12 to 17 years of age
- Assessment of changes from baseline in daily patient symptom assessment as reported by the patient.
- Assessment of changes from baseline in Physician Global Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (40):
- United States (28):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Wilmington, Delaware
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Waltham, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Plymouth, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Binghamton, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Burlington, Vermont
  - Research Site, Norfolk, Virginia
- Canada (7):
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Parkdale, Prince Edward Island
- France (3):
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Tours
- Italy (2):
  - Research Site, Genova, GE
  - Research Site, Roma, Roma

REFERENCES:
- [Derived] Gunasekaran T, Tolia V, Colletti RB, Gold BD, Traxler B, Illueca M, Crawley JA. Effects of esomeprazole treatment for gastroesophageal reflux disease on quality of life in 12- to 17-year-old adolescents: an international health outcomes study. BMC Gastroenterol. 2009 Nov 18;9:84. doi: 10.1186/1471-230X-9-84. PMID 19922626